CLINICAL TRIAL: NCT03289052
Title: A Randomized, Multi-center, Evaluator-blinded, No-treatment Controlled Study to Evaluate the Effectiveness and Safety of Restylane Volyme for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Brief Title: Restylane Volyme for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH1626
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Midface Volume Deficit
Keywords: Hyaluronic acid, midface

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Volyme (Experimental): Single injection and optional touch up injection with Restylane Volyme in Midface
  Interventions: Device: Restylane Volyme
- No intervention arm (No Intervention): No treatment

INTERVENTIONS:
Device: Restylane Volyme — Subcutis injection
  Arms: Restylane Volyme

SUMMARY:
This is a randomized, evaluator-blinded, no-treatment controlled study in subjects with Midface Volume Deficit and/or Midface Contour Deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Men or women aged 18 years of age or older of Chinese origin
3. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study
4. Subjects seeking augmentation therapy for the midface
5. MMVS score of 2, 3 or 4 on each side of the face as assessed by the blinded evaluator

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable HA gel/local anaesthetics, e.g.lidocaine or other amide-type anaesthetics.
2. Previous surgery or tattoo in the area to be treated
3. Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the lower orbital rim.
4. Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim or neurotoxin within 9 months before treatment.
5. Scars or deformities, active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema, rosacea, acne psoriasis and herpes zoster near or in the area to be treated.
6. Other condition preventing the subject from entering the study in the Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Med AB, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: The first 2 eligible subjects for each Treating Investigator will receive Restylane Volyme treatment as Group A. The injection technique will be evaluated by the Sponsor and performed after the subjects in Group A for each site have received their first treatment. If treatments are found to be correctly performed, no further training is needed, there are no outstanding questions regarding the injection technique and no other corrective actions are identified, the enrolment in Group B can start for that site. A maximum dosage of 2 mL per treatment site (i.e., right and left midface respectively) is recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively.
- Group B-Restylane Volyme Treatment Arm: Including treatment arm. A maximum dosage of 2 mL per treatment site (i.e., right and left midface respectively) is recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively.
- Group B- Control Arm: Including control arm Subjects assigned to the Control Group in Group B will not receive treatment at baseline but will return for routine follow-up for 12 months. At month 6 visit, subjects in Control Group will be offered a treatment and an optional touch-up treatment. A maximum dosage of 2 mL per treatment site (i.e., right and left midface respectively) is recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively.
Period: Overall Study
Arm/Group | Group A | Group B-Restylane Volyme Treatment Arm | Group B- Control Arm
Started | 20 | 111 | 37
Completed | 20 | 108 | 32
Not Completed | 0 | 3 | 5

BASELINE CHARACTERISTICS:
Population: All summaries will be done separately for Group A (20subjects) and B(148 subjects). For statistical inference, only Group B will be used.
Groups:
- Group A: The first 2 eligible subjects for each Treating Investigator will receive treatment as Group A.
- Restylane Volyme Treatment Group of Group B: Subjects assigned in this group will receive Restylane Volyme treatment at day 1.
- Control Group of Group B: Subjects assigned in this group will receive no treatment at day 1, but at 6m visit.
- Total: Total of all reporting groups
Arm/Group | Group A | Restylane Volyme Treatment Group of Group B | Control Group of Group B | Total
Number analyzed (Participants) | 20 | 111 | 37 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 109 | 37 | 166
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.7) | 41.3 (10.2) | 41.2 (10.0) | 41.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 104 | 32 | 156
  Male | 0 | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese Han | 20 | 111 | 37 | 168
Region of Enrollment [Number; unit: participants]
  China | 20 | 111 | 37 | 168

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: Percentage of responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face concurrently, as measured by the blinded evaluator at 6 months after last treatment in Treatment Group, and at 6 months after randomization in Control Group.
  MMVS is a Four-Point scale that assesses the fullness of the midface from Fairly Full (1) to Substantial Loss of Fullness (4) as described below. The blinded evaluator and treating investigator will rate the subject's right and left midface for severity of volume deficiency using the MMVS at all applicable study visits.
Time Frame: 6 month
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Group A: The first 2 eligible subjects for each Treating Investigator will receive Restylane Volyme treatment as Group A. The injection technique will be evaluated by the Sponsor and performed after the subjects in Group A for each site have received their first treatment. If treatments are found to be correctly performed, no further training is needed, there are no outstanding questions regarding the injection technique and no other corrective actions are identified, the enrolment in Group B can start for that site.
- Group B-treatment Arm: Subject assigned in this group will receive Restylane Volyme treatment at D1.
- Group B-control Arm: Subject assigned in this group will not receive Restylane Volyme treatment at D1 but on 6M visit.
Arm/Group | Group A | Group B-treatment Arm | Group B-control Arm
Number analyzed (Participants) | 20 | 111 | 37
percentage of subjects | 80 [56.3 to 94.3] | 87.2 [79.4 to 92.8] | 76.7 [57.7 to 90.1]

ADVERSE EVENTS:
Time Frame: 1 year.
Description: Each subject will be questioned about AEs at each clinical visit following the screening visit. The question asked will be "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination or from a laboratory test, observations by the study personnel, subject diaries or spontaneous reports from the subjects.
Groups:
- Group B-treatment Arm: including treatment arm A maximum dosage of 2 mL per treatment site (i.e., right and left midface respectively) is recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively.
- Group B-control Arm: including control arm Subjects assigned to the Control Group in Group B will not receive treatment at baseline but will return for routine follow-up for 12 months. At month 6 visit, subjects in Control Group will be offered a treatment and an optional touch-up treatment.
Arm/Group | Group A | Group B-treatment Arm | Group B-control Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/111 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/111 | 0/37
Other Adverse Events (participants affected / at risk) | 0/20 | 0/111 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=20) | Group B-treatment Arm (N=111) | Group B-control Arm (N=37)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03289052/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03289052/SAP_003.pdf